CLINICAL TRIAL: NCT00583232
Title: Protein and Energy Metabolism in Pediatric Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: GlaxoSmithKline (Industry); Crohn's and Colitis Foundation (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0506-19; IRB 0506-19
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Crohn's Disease; Protein Metabolism; Energy Metabolism
Keywords: Pediatric; Crohn's disease; protein metabolism; energy metabolism
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corticosteroid (Active Comparator): Subjects receiving corticosteroid therapy (1-2 mg/kg/day up to 60mg/day) with taper.
  Interventions: Drug: Stable isotope infusions
- infliximab (Active Comparator): Subjects receiving infliximab therapy (5 mg/kg at 0, 2 and 6 weeks, followed by every 8 week therapy)
  Interventions: Drug: Stable isotope infusions

INTERVENTIONS:
Drug: Stable isotope infusions — Stable isotope infusion will be given via an intravenous catheter. Subjects will receive a priming dose and a continuous dose.

SUMMARY:
The metabolic response to Crohn's disease, including increased proteolysis and lipolysis and changes in energy expenditure, plays a significant role in the resulting malnutrition from which these patients suffer. Tumor necrosis factor-alpha (TNF-alpha), a pro-inflammatory cytokine, has been found to be elevated in children with ulcerative colitis. TNF-alpha has been incriminated in the mechanism of weight loss in many different chronic diseases, and causes net protein and lipid catabolism. Anti-TNF-alpha antibody (infliximab) has been proven to be an effective therapy for ulcerative colitis.

The purpose of this study is to compare changes in protein and lipid metabolism, as well as resting energy expenditure, before and after therapy with anti-TNF-alpha antibody (infliximab) or corticosteroids in children with recurrent Crohn's disease. Performing this study will better define the changes in nutrition status observed in these children following remission of active Crohn's disease, and potentially lead to changes in medical and nutritional management of these children.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children between the ages of six and eighteen years of age with recurrence of active Crohn's disease, determined by their primary pediatric gastroenterologist to require either:

  1. Corticosteroid therapy ((1-2 mg/kg/d up to maximum of 60 mg/day) with taper, or
  2. Infliximab therapy (5 mg/kg at 0, 2, and 6 weeks, followed by q 8 week therapy)
* Crohn's disease of at least 3 months since diagnosis, with gastritis, duodenitis, ileitis, ileocolitis, or colitis, confirmed by endoscopy and biopsy
* PCDAI score >20
* If receiving concomitant medications, must have been on a stable regimen as follows:

  1. Subjects on aminosalicylates and/or immunomodulators should be on a stable dose for at least 2 weeks prior to enrollment.
  2. Subjects must be off oral, rectal, and parenteral corticosteroids at least 2 weeks prior to enrollment.
* Screening laboratory tests that meet the following criteria (obtained within 4 weeks of enrollment):

  1. Hemoglobin >8.0 g/dL
  2. White blood cell count >3.5 x 109/L
  3. Neutrophils >1.5 x 109/L
  4. Platelets >100 x 109/L
  5. Aspartate aminotransferase, alanine aminotransferase, and alkaline phosphatase levels within 3 times the upper limit of normal.
* For those patients to receive infliximab, PPD skin tests with skin induration <5 mm.
* Signed written consent from the parent/legal guardian and assent from the child to be obtained prior to enrollment.

Exclusion Criteria:

* Local manifestations of Crohn's disease, including fistula(s), strictures, abscesses, or other complications for which surgery may be indicated.
* Surgery for bowel diversion with placement of stoma within 3 months prior to screening.
* Positive stool examination of enteric pathogens including Salmonella and Shigella species, Clostridium difficile, and Giardia lamblia.
* Female subjects who are pregnant, nursing, or planning pregnancy.
* Concomitant diagnosis or history of congestive heart failure.
* Treatment with parenteral nutrition within 4 weeks of enrollment.
* Serious infection in the 3 months prior to enrollment.
* History of prior or current active or latent tuberculosis.
* Immune deficiency syndrome, including documented human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS).
* History of systemic lupus erythematosus.
* A transplanted organ.
* Known malignancy or history of malignancy within 5 years of enrollment.
* History of demyelinating disease.
* History of substance abuse.
* Poor tolerability of venipuncture or lack of venous access during the study period.
* A live virus vaccination within 3 months of enrollment.
* Prior history of infliximab infusion, or any other therapeutic agent targeted at reducing tumor necrosis factor-a (TNF-a).
* Hypersensitivity to any murine proteins or other component of infliximab for those patients to receive infliximab.
* Inability to comply with study procedures

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Compare whole body and splanchnic protein kinetics and balance in response to corticosteroid and anti-TNF-alpha therapies in the fasting state and during enteral nutrition infusion. | Week 0, 2 and 14

SECONDARY OUTCOMES:
Compare the effects of corticosteroid and anti-TNF-alpha therapies on resting and total energy expenditure. | Week 0, 2 and 14
Compare the effects of corticosteroid and anti-TNF-alpha therapies on free fatty acid metabolism | Week 0, 2 and 14
Compare the effects of corticosteroid and anti-TNF-alpha therapies on quality of life | Week 0, 2, and 14
Comparing the effects of corticosteroid and anti-TNF-alpha therapies on bone turnover and bone density | Week 0,2 and 14
Compare the effects of corticosteroid and anti-TNF-alpha therapies on body composition. | Week 0, 2 and 14
Compare the effects of corticosteroid and anti-TNF-alpha therapies on cytokines known to be altered in inflammatory bowel disease. | Week 0, 2 and 14
Compare the effects of corticosteroid and anti-TNF-alpha therapies on vascular endothelial function. | Week 0, 2 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Steiner, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University-Riley Hospital for Children, Indianapolis, Indiana, United States